CLINICAL TRIAL: NCT01090817
Title: A Multicentre Australian Phase 2 Study to Evaluate Safety and Efficacy of Mesenchymal Stromal Cells for Treating Biologic Refractory Crohn's Disease
Brief Title: An Australian Study of Mesenchymal Stromal Cells for Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R.P.Herrmann (Other)
Collaborators: The Queen Elizabeth Hospital (Other); Concord Hospital (Other); Sir Charles Gairdner Hospital (Other); The Alfred (Other)
Responsible Party: Sponsor-Investigator, R.P.Herrmann, Director Cell and Tissue Therapies Western Australia, Royal Perth Hospital
Organization: Royal Perth Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC2009/123; CTN2010/0098 (Other: Therapeutics Good Administration, Government of Australia)
Record Dates: First submitted 2010-03-22; First posted 2010-03-23 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Crohn Disease
Keywords: mesenchymal stromal cells; ileitis; colitis
MeSH Terms: conditions — Crohn Disease; Ileitis; Colitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal stromal cells (Experimental): Mesenchymal stromal cells administered weekly for 4 weeks
  Interventions: Drug: Mesenchymal stromal cells (MSC) for infusion

INTERVENTIONS:
Drug: Mesenchymal stromal cells (MSC) for infusion — MSC 2X10E6/kg recipient weight are infused over 15 minutes intravenously weekly for 4 weeks
  Other Names: No other names

SUMMARY:
Despite the advent of newer biologic therapies such as infliximab for Crohn's disease, a form of autoimmune inflammatory bowel disease, a proportion of patients are refractory to such therapy and require surgery. The hypothesis is that mesenchymal stromal cell therapy using third party human cultured cells will be safe and effective

ELIGIBILITY:
Inclusion Criteria:

* Colonic or small bowel Crohn's disease based on endoscopic appearances and histology
* Refractory to induction with infliximab or adalimumab; or have lost response to these agents; or have had side effects precluding their further use
* Where there has been loss of response to one of these agents, the other must be tried before being eligible
* Crohn's disease activity score (CDAI) 250 or more.
* C-reactive protein >10mg/L
* Surgery must have been offered to the subject (if appropriate) and declined
* Signed informed consent

Exclusion Criteria:

* Active sepsis, perforating disease. Coexistent perianal fistulous disease is permitted, providing no co-existent infection within previous 4 weeks
* Chronic stricturing disease in isolation
* Coexistent CMV disease
* Prior history of malignancy
* Pregnant or unwilling to practice contraceptive therapy or breast feeding females
* Last biologic therapy must be greater than 4 weeks prior, must be on stable corticosteroid dose for 14 days prior, during therapy and for 14 days after therapy, must be on stable immunomodulator dose (eg, azathioprine) for 14 days prior, during therapy and for 14 days after.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-01; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Clinical response to MSC: Reduction of Crohn's disease Activity score by 100 points or more at six weeks post start of therapy | Six weeks
  Colonoscopy and biopsy as well as clinical parameters used for the Crohn's disease acivity (www.ibdaustralia.org/cdai/) will be undertaken at screening pre-therapy and at 6 weeks after start of therapy.

SECONDARY OUTCOMES:
Incidence of infusional toxicity | Six weeks
  Subjects will receive mesenchymal stromal cell therapy, 2X10E6/kg weekly by IV infusion for 4 weeks and will be assessed for 4 hours post infusion
Induction of remission | Six weeks
  Crohn's disease activity index assessed as below 150
Improved quality of life | Six weeks
  Increase in IBDQ and SF-36 scores measured at six weeks
Endoscopic improvement. | Six weeks
  Crohn's disease endoscopic improvement score will be measured at repeat endoscopy six weeks after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Forbes, MD, Principal Investigator — Royal Perth Hospital
Locations (1):
- Department of Gastroenterology and Hepatology, Royal Perth Hospital, Perth, Western Australia, Australia

REFERENCES:
- [Derived] Forbes GM, Sturm MJ, Leong RW, Sparrow MP, Segarajasingam D, Cummins AG, Phillips M, Herrmann RP. A phase 2 study of allogeneic mesenchymal stromal cells for luminal Crohn's disease refractory to biologic therapy. Clin Gastroenterol Hepatol. 2014 Jan;12(1):64-71. doi: 10.1016/j.cgh.2013.06.021. Epub 2013 Jul 19. PMID 23872668